CLINICAL TRIAL: NCT01072136
Title: A Randomized Trial to Evaluate the Need for Empiric Therapy for Mucopurulent Cervicitis of Unknown Etiology
Brief Title: Empiric Therapy of Mucopurulent Cervicitis (MPC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07-0082
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2012-01

CONDITIONS: Vaginitis Bacterial; Cervicitis
Keywords: mucopurulent cervicitis, chlamydia, gonorrhea, women
MeSH Terms: conditions — Vaginosis, Bacterial; Uterine Cervicitis; Chlamydia Infections; Gonorrhea | interventions — Azithromycin; Cefixime

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator): Placebo.
  Interventions: Other: Placebo
- Azithromycin/Cefixime (Experimental): A single dose of cefixime 400 mg (1 tablet oral at 400 mg) and azithromycin 1 gram (2 tablets oral at 500 mg each).
  Interventions: Drug: Azithromycin; Drug: Cefixime

INTERVENTIONS:
Other: Placebo — Capsule will be filled with lactose and be identical in appearance to the capsule with the active ingredient.
  Arms: Placebo
Drug: Azithromycin — Single dose will consist of 2 over-encapsulated capsules (500 mg each) administered orally.
  Arms: Azithromycin/Cefixime
Drug: Cefixime — Single dose will consist of 1 over-encapsulated capsule (400 mg) administered orally.
  Arms: Azithromycin/Cefixime

SUMMARY:
Mucopurulent cervicitis (MPC) is a syndrome with associated symptoms including mucopurulent discharge (mucus and pus) from the cervix and other signs of inflammation such as easily induced cervical bleeding. The purpose of this study is to evaluate the effectiveness of no treatment versus empiric treatment with a single dose of cefixime and azithromycin for cure of MPC. Empiric treatment is the initiation of treatment prior to a firm diagnosis. Study participants will include 772 women ages 18 and older in good health with MPC. Women will be randomly assigned to 1 of 2 possible study groups: Group 1 will receive a single dose of cefixime and azithromycin antibiotics and Group 2 will receive placebo (inactive substance). Study procedures will include pelvic examination with a cervical swab sample. Participants will be involved in study related procedures for approximately 2 months, which includes 3 study visits.

DETAILED DESCRIPTION:
Mucopurulent cervicitis (MPC) is a clinical syndrome characterized by the presence of mucopurulent discharge from the cervix and other signs of inflammation such as easily induced cervical bleeding. This phase III study is designed to evaluate the effectiveness of no treatment (placebo) versus empiric treatment with a single dose of cefixime 400 mg and azithromycin 1 gram for clinical cure of MPC at 2 months of follow-up. Secondary aims of the study are: to compare the pelvic inflammatory disease (PID) rate and adverse event rates between no treatment (placebo) versus empiric treatment; explore the role of bacterial vaginosis and Mycoplasma genitalium in the persistence of MPC; evaluate microbiological cure rate of M. genitalium in women treated with cefixime and azithromycin versus placebo; and present the clinical cure, partial response and failure proportions at 2-3 weeks and 2 months for each study arm. Participants will include 772 women greater than or equal to 18 years of age from Sexually Transmitted Disease (STD) or Family Planning (FP) clinics in good general health with MPC in New Orleans, LA; Birmingham, AL; Jackson, MS; Los Angeles, CA; and an additional site to be determined. Research specimens will be obtained at the time of the pelvic examination. As part of the study protocol, 3 cervical and 4 vaginal swabs will be collected at screening, follow-up visit 1, and follow-up visit 2. Eligible participants with clinical MPC at the time of their pelvic examination (cervical mucopus or easily induced cervical bleeding), will be consented, screened, enrolled, and randomized to one of the following arms: Group 1: empiric treatment: a single dose of cefixime 400 mg (1 capsule oral at 400 mg) and azithromycin 1 gm (2 capsules oral at 500 mg each) or Group 2: no treatment: placebo pills that look identical to the above medications. Subjects will be involved in study related procedures for 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Women greater than or equal to 18 years old in Sexually Transmitted Disease (STD) clinics or Family Planning clinics.
* Presence of cervical mucopus and/or easily induced cervical bleeding on pelvic exam via endocervical swab.
* Greater than or equal to 30 white blood cells (WBCs) per high power field in the cervical Gram stain. (Note: the cervical Gram stains will be sent to a central lab for review. The results will not be available at the time of enrollment. Subjects who do not meet this criterion will be withdrawn from the study at the time the results are available).
* Willingness to provide written informed consent
* Willing to abstain from sexual intercourse or use condoms during the entire study (approximately 2 months).
* Willing to abstain from using vaginal products during the entire study (approximately 2 months).

Exclusion Criteria:

* Signs and symptoms of pelvic inflammatory disease, including cervical motion, uterine, or adnexal tenderness.
* History of pelvic inflammatory disease (PID), ectopic pregnancy or recurrent cervicitis (3 or more episodes in the prior year) or written documentation of recent cervicitis (within past 30 days).
* Gonorrhea or Chlamydia on nucleic acid amplification test (NAAT) at time of enrollment. (Participant testing positive for Neisseria gonorrhoeae (GC) or Chlamydia trachomatis (CT) on enrollment visit sample will be discontinued).
* Women with motile trichomonas on wet mount examination or positive trichomonas culture at time of enrollment.
* Women with symptomatic bacterial vaginosis (BV) (based on clinical Amsel criteria for BV and reported symptoms by participant, i.e. discharge, vaginal odor, etc).
* Use of vaginal products in past 48 hours (i.e. douching, use of vaginal medications or suppositories).
* History of chronic renal disease by verbal or documented history.
* Current use of probenecid.
* Nursing mothers.
* Colitis or coagulopathy as per patient self-report.
* Known allergy to cephalosporins, penicillin or macrolides by verbal or documented history.
* History of latex allergy.
* Use of systemic antibiotics (oral or intravenous), vaginal antibiotics, vaginal antifungal, or oral antifungal use within 30 days of study enrollment.
* Women who will require antibiotic treatment due to GC or CT in a sexual partner.
* Serious underlying conditions, including human immunodeficiency virus (HIV) or other primary or secondary immunosuppressive condition.
* Concomitant infection, which requires antimicrobial therapy (for example, urinary tract infection, sinusitis, skin and soft tissue infection, tooth abscess, etc.) or expected use of any antibiotic/antimicrobial therapy during the study.
* Menstruation at the time of screening visit. Women who are menstruating can be screened after cessation of bleeding.
* Active herpes outbreak at the time of enrollment determined by clinical observation.
* Suspected pregnancy or positive urine pregnancy test at screening or actively seeking pregnancy during study period.
* Any clinical adverse event, intercurrent illness, or other medical condition or situation as determined by the investigator that is present or occurs such that participation in the study would not be in the best interest of the participant.
* Previously enrolled in this study.
* Unable to follow the protocol (inc. inability to comply with the follow-up procedures).
* Failing to provide contact information.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-03; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Alabama Hospital - Infectious Diseases, Birmingham, Alabama
  - Harbor UCLA Medical Center - OBGYN - General Gynecology and Women's Health, Torrance, California
  - Louisiana Stte University - Health Sciences Center - Medicine, New Orleans, Louisiana
  - University of Mississippi - Infectious Diseases, Jackson, Mississippi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from STD or family planning clinics in New Orleans, LA, Birmingham AL, Jackson, MS, and Los Angeles CA between March 2010 and May 2011.
Period: Overall Study
Arm/Group | Azithromycin/Cefixime | Placebo
Started | 44 | 43
Met All Enrollment Criteria | 30 (Some eligibility test results were not available until after randomization.) | 25
Completed | 21 | 12
Not Completed | 23 | 31

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin/Cefixime | Placebo | Total
Number analyzed (Participants) | 30 | 25 | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 25 | 55
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (6.6) | 25.8 (6.3) | 25.8 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 25 | 55

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Clinical Cure in Participants Not Treated Versus Participants Empirically Treated With Cefixime and Azithromycin for Mucopurulent Cervicitis (MPC).
Description: The proportion of participants who have cleared MPC by the second follow-up visit. Clinical cure is defined as: absence of cervical mucopus and absence of easily induced cervical bleeding and < 30 white blood cells per oil immersion field on cervical gram stain.
Time Frame: Visit 2 - 2 months (Day 50-70).
Population: Per protocol. Received study product, met eligibility criteria, had complete primary outcome data, and absence of any major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin/Cefixime | Placebo
Number analyzed (Participants) | 21 | 12
percentage of participants | 19 | 33
Statistical Analysis 1: Comparison: Azithromycin/Cefixime vs Placebo; The primary efficacy outcome was MPC clinical cure at 2 months. This was a non-inferiority trial designed to reject the null hypothesis that placebo control is inferior to empiric therapy for MPC; Test type: Non-Inferiority or Equivalence — Under the assumption of a clinical cure proportion of 75% for the Azithromycin/Cefixime group, a 10% non-inferiority margin (i.e., no more than a 10% lower cure rate in the placebo group) at the one-sided 0.05 significance level with 85% power required 270 study participants in each arm (540 total) using an unpooled Z-test (normal approximation). Anticipating that approximately 30% of enrolled participants would not be in the per protocol group, 772 participants were targeted for enrollment; Risk Difference (RD) = 14.0, 95% CI 1-sided [lower limit -12.2] — Asymptotic one-sided 95% confidence limit for the difference in clinical cure proportions(placebo minus treatment) were computed so that the lower limit could be examined relative to the non-inferiority margin of -10%

2. Secondary Outcome: Determine Pelvic Inflammatory Disease (PID) in Patients Empirically Treated With Cefixime and Azithromycin for Mucopurulent Cervicitis (MPC) in Comparison to no Treatment.
Description: The number of participants experiencing PID after randomization.
Time Frame: At 2-3 week and 2 month (Day 50-70) follow-up.
Population: Participants who were randomized and received study product.
Measure: Number; unit: participants
Arm/Group | Azithromycin/Cefixime | Placebo
Number analyzed (Participants) | 44 | 43
participants | 1 | 0

3. Secondary Outcome: Examine Adverse Events in Patients Empirically Treated With Cefixime and Azithromycin for Mucopurulent Cervicitis (MPC) in Comparison to no Treatment.
Description: The proportion of participants experiencing one or more adverse events after randomization.
Time Frame: At 2-3 week and 2 month (Day 50-70) follow-up.
Population: Participants who were randomized and received study product.
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin/Cefixime | Placebo
Number analyzed (Participants) | 44 | 43
percentage of participants | 36.4 | 27.9

4. Secondary Outcome: Explore the Role of Bacterial Vaginosis (BV) in Persistent Mucopurulent Cervicitis (MPC).
Description: Proportion of participants with clinical failure, partial response, or clinical cure for mucopurulent cervicitis at 2 month follow-up according to asymptomatic bacterial vaginosis status at 2 month follow-up.
  Clinical Failure:
  * Persistent cervical mucopus and/or easily induced cervical bleeding, and the presence of > 30 WBCs per oil immersion field on cervical gram stain OR
  * Signs of pelvic inflammatory disease, including cervical motion tenderness, uterine tenderness or adnexal tenderness.
  Partial Response:
  * Persistent cervical mucopus and/or easily induced cervical bleeding and <30 WBCs per oil immersion field on cervical gram stain OR
  * The presence of ≥ 30 WBCs per oil immersion field on cervical gram stain in the absence of both cervical mucopus and easily induced cervical bleeding.
  Clinical Cure:
  • Absence of cervical mucopus and absence of easily induced cervical bleeding and < 30 WBC's per oil immersion field on cervical gram stain.
Time Frame: At 2 month (Day 50-70) follow-up.
Population: Participants who met eligibility criteria and were not positive for chlamydia, gonorrhea, cervical trichomonas or cervical mycoplasma genitalium at 2 month follow-up.
Measure: Number; unit: percentage of participants
Groups:
- Clinical Failure: Clinical failure for mucopurulent cervicitis
- Partial Response: Partial response for mucopurulent cervicitis
- Clinical Cure: Clinical Cure for mucopurulent cervicitis
Arm/Group | Clinical Failure | Partial Response | Clinical Cure
Number analyzed (Participants) | 9 | 16 | 7
percentage of participants
  No Asymptomatic Bacterial Vaginosis | 78 | 88 | 43
  Asymptomatic Bacterial Vaginosis | 22 | 13 | 57

5. Secondary Outcome: Explore the Role of Mycoplasma Genitalium in Persistent Mucopurulent Cervicitis (MPC).
Description: Proportion of participants with clinical failure, partial response, or clinical cure for mucopurulent cervicitis at 2 months according to mycoplasma genitalium status(positive cervical or vaginal swabs versus both negative) at 2 months.
  Clinical Failure:
  * Persistent cervical mucopus and/or easily induced cervical bleeding, and the presence of > 30 WBCs per oil immersion field on cervical gram stain OR
  * Signs of pelvic inflammatory disease, including cervical motion tenderness, uterine tenderness or adnexal tenderness.
  Partial Response:
  * Persistent cervical mucopus and/or easily induced cervical bleeding and <30 WBCs per oil immersion field on cervical gram stain OR
  * The presence of ≥ 30 WBCs per oil immersion field on cervical gram stain in the absence of both cervical mucopus and easily induced cervical bleeding.
  Clinical Cure:
  • Absence of cervical mucopus and absence of easily induced cervical bleeding and < 30 WBC's per oil immersion field on cervical gram stain.
Time Frame: At 2 month (Day 50-70) follow-up.
Population: Participants who met eligibility criteria and were not positive for chlamydia, gonorrhea, cervical trichomonas at 2-month follow-up.
Measure: Number; unit: percentage of participants
Arm/Group | Clinical Failure | Partial Response | Clinical Cure
Number analyzed (Participants) | 9 | 16 | 7
percentage of participants
  Negative for mycoplasma genitalium | 100 | 94 | 100
  Positive for mycoplasma genitalium | 0 | 6 | 0

6. Secondary Outcome: Evaluate Microbiological Cure of Mycoplasma Genitalium in Women Treated With Cefixime and Azithromycin Versus Placebo.
Description: The proportion of participants with mycoplasma genitalium at baseline who clear mycoplasma genitalium in either the vagina or cervix at their last follow-up visit.
Time Frame: At 2-3 weeks and 2 month (Day 50-70) follow-up.
Population: Participants who were positive for mycoplasma genitalium in either the cervix or vagina at baseline and who met eligibility criteria and who returned for at least one of the follow-up visits.
Measure: Number; unit: participants
Arm/Group | Azithromycin/Cefixime | Placebo
Number analyzed (Participants) | 4 | 3
participants | 2 | 1

7. Secondary Outcome: Determine the Clinical Cure, Partial Response and Failure Proportions for Mucopurulent Cervicitis at 2 Months for Each Study Arm.
Description: Clinical Failure:
  * Persistent cervical mucopus and/or easily induced cervical bleeding, and the presence of > 30 WBCs per oil immersion field on cervical gram stain OR
  * Signs of pelvic inflammatory disease, including cervical motion tenderness, uterine tenderness or adnexal tenderness.
  Partial Response:
  * Persistent cervical mucopus and/or easily induced cervical bleeding and <30 WBCs per oil immersion field on cervical gram stain OR
  * The presence of ≥ 30 WBCs per oil immersion field on cervical gram stain in the absence of both cervical mucopus and easily induced cervical bleeding.
  Clinical Cure:
  • Absence of cervical mucopus and absence of easily induced cervical bleeding and < 30 WBC's per oil immersion field on cervical gram stain.
Time Frame: At 2 month ( Day 50-70) follow-up.
Population: Per protocol. Received study product, met all eligibility criteria, had complete primary outcome data, and absence of any major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin/Cefixime | Placebo
Number analyzed (Participants) | 21 | 12
percentage of participants
  Clinical cure | 19 | 33
  Partial response | 43 | 50
  Clinical failure | 38 | 17

8. Secondary Outcome: Determine the Clinical Cure, Partial Response and Failure Proportions for Mucopurulent Cervicitis at 2-3 Weeks for Each Study Arm.
Description: as for outcome 7
Time Frame: At 2-3 weeks follow-up.
Population: Received study product, met all eligibility criteria, and had complete outcome data at 2-3 weeks.
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin/Cefixime | Placebo
Number analyzed (Participants) | 27 | 18
percentage of participants
  Clinical cure | 7 | 0
  Partial response | 41 | 72
  Clinical failure | 52 | 28

ADVERSE EVENTS:
Arm/Group | Azithromycin/Cefixime | Placebo
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/43
Other Adverse Events (participants affected / at risk) | 11/44 | 1/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Azithromycin/Cefixime (N=44) | Placebo (N=43)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)

LIMITATIONS AND CAVEATS:
The study closed early due to slow accrual with 11% of the targeted sample size enrolled. Therefore, precision and power were low.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No